CLINICAL TRIAL: NCT02562820
Title: Ketamine for the Treatment of Rett Syndrome: An Exploratory Trial
Brief Title: An Exploratory Trial of Ketamine for the Treatment of Rett Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-627
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Subjects will receive intravenous infusion of a 0.1, 0.5, 1.0, 2.0 or 4.5 mg/kg dose over the course of 40 minutes
  Interventions: Procedure: Intravenous infusion
- Placebo (Placebo Comparator): Subjects will receive an intravenous infusion of normal saline over the course of 40 minutes
  Interventions: Procedure: Intravenous infusion

INTERVENTIONS:
Procedure: Intravenous infusion — Intravenous infusion of Ketamine
  Arms: Ketamine
Procedure: Intravenous infusion — Intravenous infusion of Normal Saline
  Arms: Placebo

SUMMARY:
Rett Syndrome (RTT) is a complex disorder resulting from mutations in a gene encoding the MeCP2 protein. Currently, there are no methods to fix the abnormal gene, however, animal studies suggest that the symptoms of RTT can be treated.

Ketamine is a sedative or anesthetic, depending on the dose. The drug is approved by the US Food and Drug Administration (FDA) and is commonly used in children and adults. Animal studies and case reports in humans suggest that ketamine may reduce the symptoms of Rett syndrome. The purpose of this study is to determine the safety and efficacy of ketamine for treating breathing and behavioral symptoms of RTT.

DETAILED DESCRIPTION:
Families will be asked to maintain current prescription medications during the expected three-month duration of the study. However, clinically indicated medication alterations will naturally be permitted and recorded.

Each participant will experience four study days, separated by about a month. On three of the study days participants will be given Ketamine, and on the other day they will be given saline placebo.

Studies will be conducted in the Cleveland Clinic's General Clinical Research Unit which is an NIH-sponsored unit designed for studies such as this. Subjects will be admitted on the first day of each study sequence, and discharged the subsequent day. Study subjects will arrive at approximately 8:00 AM. Age, weight and height will be determined and prescription medications will be recorded. Subjects will be fitted with sensors for recording respiration, heart rate and brain electrical activity (electroencephalogram, or EEG). Treatment administration will start at noon. To avoid potential effects of circadian variation, treatment administration will start at the same time for each study day in each subject. Because the half-life of Ketamine is short (t1/2 = 10-15 minutes for sedation/anesthesia), we expect participating patients to be fully recovered from any potential sedating effects of Ketamine within an hour or two.

Each subject will be randomized to receive 3 of the 5 doses of Ketamine 0.1, 0.5, 1.0, 2.0 or 4.5 mg/kg] plus placebo, for a total of 4 periods (visits). Ordering of the treatments will be randomized, with patients earlier in the study to receive lower doses of Ketamine.

The study drug will be given as a constant infusion at 0.1, 0.5, 1.0, 2.0 or 4.5 mg/kg over the course of 40 minutes.

Apnea/breath-hold index, hyperventilation and cardio-respiratory coupling indices will be measured by polysomnography (PSG) before, during and after each treatment.

EEG will be recorded before, during and after each treatment.

Auditory evoked potentials (AEP) will be recorded on the day after each treatment.

Rett Syndrome Behavior Questionnaire (RSBQ) will be administered multiple times after each treatment, first in the hospital and then at home.

Repetitive Behavior Scale-Revised (RBSR) will be administered on the day after each treatment.

Before infusion and one hour after infusion, a few mL of peripheral blood will be sampled to measure bio-markers. Blood will be centrifuged and plasma will be frozen for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Rett syndrome diagnosis based on the 2010 RTT diagnostic criteria, as determined by review of clinical records, and
2. Pathogenic mutation in the MECP2 gene, and
3. Breathing score of 3 or greater on RSBQ, and
4. Age 5-25 years.

Exclusion Criteria:

1. Ongoing clinical regression as determined by review of clinical records and consultation with parents, or
2. Seizure within one week of study session, or
3. Unstable systemic illness other than Rett syndrome, or
4. Clinically important variations in medication use.

Ages: 5 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Behavioral phenomena requiring intervention | From time of admission until time of discharge during any particular study visit, typically within 36 hours of admission.
  Occurrence of agitation, irritability, or worsening of pre-existing symptoms.

SECONDARY OUTCOMES:
Exploratory - Rett Syndrome Behavior Questionnaire (RSBQ) | On the day following study drug infusion at each visit (30 - 36 hours after admission for each visit).
  A formal score obtained by administering the RSBQ to the subject's parent/guardian before and after every study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States